CLINICAL TRIAL: NCT01414725
Title: Core Stability Training in Ambulant Individuals With Multiple Sclerosis: a Multi-centre Randomised Controlled Trial.
Brief Title: Core Stability Training in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Plymouth (Other)
Responsible Party: Principal Investigator, Jenny Freeman, Dr Jenny Freeman, University of Plymouth
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 10/H0106/88
Record Dates: First submitted 2011-08-05; First posted 2011-08-11 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2014-03

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Mobility; Balance; Core Stability; Physiotherapy
MeSH Terms: conditions — Multiple Sclerosis | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Core Stability Training (Experimental)
  Interventions: Other: Core Stability Training
- Relaxation (Placebo Comparator)
  Interventions: Other: Relaxation
- Standard Physiotherapy Exercises (Active Comparator)
  Interventions: Other: Standard Physiotherapy Exercises

INTERVENTIONS:
Other: Standard Physiotherapy Exercises — Individualised face to face training sessions, delivered over 12 weeks, plus an individualised 15-minute daily home exercise programme will be provided. This will be undertaken by a neurological physiotherapist. The exercises will comprise a standardised programme of simple physiotherapy exercises which aim to improve trunk and pelvic stability, lower limb muscle length and strength, and balance and control of movement, as described by Barrett et al [2009]. Exercises will be progressed in response to the abilities of the individual. Each participant will receive a workbook with written and diagrammatic instructions describing their home exercise programme.
  Other Names: Physiotherapy
  Arms: Standard Physiotherapy Exercises
Other: Core Stability Training — Individualised face to face training sessions, delivered over 12 weeks, plus an individualised 15-minute daily home exercise programme will be provided. This will be undertaken by a neurological physiotherapist with experience in the delivery of core stability training to people with MS. Exercises will be progressed in response to the abilities of the individual. Each participant will receive a workbook with written and diagrammatic instructions describing their home exercise programme.
  Other Names: Physiotherapy
  Arms: Core Stability Training
Other: Relaxation — Three face to face individualised relaxation sessions, provided at 4 weekly intervals, plus a 15-minute home programme based around an audio relaxation CD. Weekly telephone contact / support will be provided.
  Other Names: Physiotherapy
  Arms: Relaxation

SUMMARY:
The primary purpose of this study is to determine whether a 12 week Pilates based core stability training programme is effective in improving balance, mobility and balance confidence in ambulant individuals with Multiple Sclerosis (MS).

DETAILED DESCRIPTION:
The primary purpose of this study is to determine whether a 12 week Pilates based core stability training programme is effective in improving balance, mobility and balance confidence in ambulant individuals with Multiple Sclerosis (MS). The secondary aim is to determine the relative effectiveness of this 12 week Pilates based core stability training programme compared to a standardised physiotherapy exercise programme. Finally we intend to explore the underlying mechanisms of change associated with these exercise interventions by directly measuring changes in muscle thickness and activation in the deep abdominal core stabilising muscles of a sub-set of participants.

ELIGIBILITY:
Inclusion Criteria:

* Definite diagnosis of MS, according to McDonald's criteria
* Aged 18 years or over
* Able to walk independently with or without use of intermittent or constant unilateral assistance such as walking stick or orthotic brace

Exclusion Criteria:

* In relapse or relapse in previous three months
* Any medical condition contra-indicating participation in core stability exercises
* Score < 6 on the Abbreviated Mental Test, as an indicator of those whose cognitive difficulties could interfere with the informed consent process, or the ability to fully engage in the exercise programme.
* Current or recent (within past 6 months) participation in core stability exercises
* Current involvement in another interventional research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change in 10 metre timed walk (10MTW) | baseline (pre intervention), 12 weeks (immediately post intervention), 16 weeks ( one month follow-up)

SECONDARY OUTCOMES:
Change in Functional Reach - forwards and lateral | baseline (pre intervention), 12 weeks (immediately post intervention), 16 weeks ( one month follow-up)
Change in Visual Analogue Scale (10 point) to determine "Difficulty in carrying a drink when walking". | baseline (pre intervention), 12 weeks (immediately post intervention), 16 weeks ( one month follow-up)
Change in Activities-specific Balance Confidence (ABC) Scale | baseline (pre intervention), 12 weeks (immediately post intervention), 16 weeks (one month follow-up)
Change in Multiple Sclerosis 12-item Walking Scale | baseline (pre intervention), 12 weeks (immediately post intervention), 16 weeks (one month follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Freeman, Principal Investigator — University of Plymouth
Locations (7):
- United Kingdom (7):
  - Merlin Centre, Bradbury House, Hewas water, St Austell, Cornwall
  - Devon NHS Trust, Newton Abbot, Devon
  - University Of Plymouth, School of Health Professions, Plymouth, Devon
  - Tavistock Community Hospital, Spring Hill, Tavistock, Devon
  - Lanarkshire NHS Trust, Cumbernauld, North Lanarkshire
  - South Tees NHS Trust, Middlesbrough, South Tees
  - University College London Hospital Trust, London

REFERENCES:
- [Background] Freeman JA, Gear M, Pauli A, Cowan P, Finnigan C, Hunter H, Mobberley C, Nock A, Sims R, Thain J. The effect of core stability training on balance and mobility in ambulant individuals with multiple sclerosis: a multi-centre series of single case studies. Mult Scler. 2010 Nov;16(11):1377-84. doi: 10.1177/1352458510378126. Epub 2010 Aug 10. PMID 20699285
- [Background] Freeman J, Fox E, Gear M, Hough A. Pilates based core stability training in ambulant individuals with multiple sclerosis: protocol for a multi-centre randomised controlled trial. BMC Neurol. 2012 Apr 5;12:19. doi: 10.1186/1471-2377-12-19. PMID 22480437
- [Background] Fox et al. (2013) Pilates based core stability training in ambulant individuals with multiple sclerosis: a multicentre, blinded, randomised, placebo controlled trial Way Ahead 2014;18(1):6-8 http://www.mstrust.org.uk/professionals/information/wayahead/articles/18012014_03.jsp